CLINICAL TRIAL: NCT07397962
Title: Treatment of Histamine Intolerance Using Probiotic Intervention - a Randomized Controlled Trial in Adults With Clinical Signs of Histamine Intolerance
Brief Title: Treatment of Histamine Intolerance Using Probiotic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Lactopia GmbH, An der Römerbrücke 16, 66121 Saarbrücken, Germany (Unknown)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, MD, Professor, University of Hohenheim
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKES-HistaProbi-2023
Record Dates: First submitted 2026-01-23; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Histamin Intolerance
Keywords: Probiotics; Digestive symptoms; gut health; microbiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive Probio Histamed® (Lactopia GmbH), a multi-species probiotic preparation containing Bifidobacterium breve, Bifidobacterium lactis, Bifidobacterium infantis, Bifidobacterium longum, Lactobacillus gasseri, and Lactobacillus rhamnosus (total dose 5 × 10⁹ CFU per day).
  The product is administered as a powder (2 g per day) dissolved in a cold or warm beverage and taken once daily before a meal for four weeks.
  Interventions: Dietary Supplement: Probio Histamed®, a multi-species probiotic preparation containing Bifid. breve, Bifid. lactis, Bifid. infantis, Bifid. longum, Lact. gasseri, and Lact. rhamnosus (5 x 10⁹ CFU per day)
- Control (Placebo Comparator): Participants receive a placebo powder containing maltodextrin, identical in appearance and administration to the probiotic product.
  The placebo is administered as 2 g per day dissolved in a cold or warm beverage and taken once daily before a meal for four weeks.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Dietary Supplement: Probio Histamed®, a multi-species probiotic preparation containing Bifid. breve, Bifid. lactis, Bifid. infantis, Bifid. longum, Lact. gasseri, and Lact. rhamnosus (5 x 10⁹ CFU per day) — Multi-species probiotic preparation containing Bifidobacterium breve, Bifidobacterium lactis, Bifidobacterium infantis, Bifidobacterium longum, Lactobacillus gasseri, and Lactobacillus rhamnosus (total dose 5 × 10⁹ CFU per day).
  The product is administered as a powder (2 g per day) dissolved in a cold or warm beverage and taken once daily before a meal for four weeks.
  Arms: Intervention
Other: Placebo Control — maltodextrin
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if a probiotic product can lower symptoms in adults with histamine intolerance. Histamine intolerance can cause stomach and bowel problems as well as symptoms such as flushing, itching, headaches, and dizziness. The study will also learn how safe and well tolerated the probiotic is.

The main questions this study aims to answer are:

Does the probiotic lower digestive symptoms linked to histamine intolerance?

Does it lower other common symptoms, such as flushing, itching, headaches, or dizziness?

Researchers will compare the probiotic to a placebo. A placebo is a look-alike powder that contains no active bacteria. This will help determine whether the probiotic works better than no treatment.

Participants will:

Take either the probiotic or the placebo once a day for four weeks

Visit the study center for screening and two study visits

Answer symptom questionnaires

Provide blood samples and urine samples

The study is for adults with symptoms of histamine intolerance. Participation is voluntary, and participants can stop taking part at any time.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Symptoms of histamine intolerance (based on medical history)
* DAO < 10 U/mL
* Age 18-70 years
* Willingness to refrain from changing eating habits and physical activity during the study
* Sufficient understanding of the German language and sufficient mental state to understand information and instructions related to the study

Exclusion Criteria:

* Lactose intolerance
* Fructose malabsorption
* Helicobacter pylori infection
* Celiac disease
* Chronic inflammatory bowel disease
* Food allergy with gastrointestinal manifestation
* Mastocytosis
* Use of antihistamines
* Other gastrointestinal diseases or use of gastrointestinal medications, as determined by the investigator
* (Planned) change in current medication, as determined by the investigator
* Pregnancy and breastfeeding
* Inability to take the investigational drug orally
* Intolerance to the investigational drug
* Admission to a clinic or similar facility due to official or court order
* Participation in another clinical trial (currently or within the last 30 days prior to study start)
* A health condition or regular medication use that, in the opinion of the investigator, does not allow participation in the study or the evaluation of study parameters or the consumption of the investigational drug (individual decision)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Irritable bowel severity scoring system (IBS-SSS) | From baseline to the end of the study (4 weeks)
  Chang of total score of IBS-SSS, a score ranging from 0 to 500. High values mean high gastrointestinal symptoms.

SECONDARY OUTCOMES:
Facial flushing | From baseline to the end of the study (4 weeks)
  Facial flushing is measured on a visual analogue scale ranging from 0 to 100 with higher values meaning more pronounced symptoms.
Itching | From baseline to the end of the study (4 weeks)
  Itching is measured on a visual analogue scale ranging from 0 to 100 with higher values meaning more pronounced symptoms.
Headache | From baseline to the end of the study (4 weeks)
  Headache is measured on a visual analogue scale ranging from 0 to 100 with higher values meaning more pronounced symptoms.
Dizziness | From baseline to the end of the study (4 weeks)
  Dizziness is measured on a visual analogue scale ranging from 0 to 100 with higher values meaning more pronounced symptoms.

OTHER OUTCOMES:
Concentration of Diaminooxidase in capillary blood | From baseline to the end of the study (4 weeks)
Concentration of Methylhistamine in urine | From baseline to the end of the study (4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für klinische Ernährung Stuttgart, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No